CLINICAL TRIAL: NCT04867460
Title: Ultrasound-guided Venous Access, Using a Wireless Probe, for Pacemaker and Defibrillator Implants - a Randomized Study
Brief Title: Ultrasound-guided Venous Access for Pacemaker and Defibrillator Implants
Acronym: TUFF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment too slow. Unrealistic to finish study with full recruitment.
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TUFF-study
Record Dates: First submitted 2021-04-27; First posted 2021-04-30 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2024-04

CONDITIONS: Cardiac Arrhythmia; Heart Failure; AV Block
Keywords: Pacemaker; Implantable defibrillator; Venous access; Ultrasound
MeSH Terms: conditions — Arrhythmias, Cardiac; Heart Failure; Atrioventricular Block

STUDY DESIGN:
Intervention Model Description: 1:1 randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound guided venous access (Experimental): Vascular access of the axillary vein will be performed using an ultrasound system (Siemens Acuson Freestyle) with a wireless vascular ultrasound probe (L8-3 or L13-5). One or more vascular punctures will be performed, as needed.
  Interventions: Procedure: Ultrasound guided venous access
- Standard of care (No Intervention): Vascular access of the axillary or subclavian vein will be performed using anatomical landmarks, fluoroscopy and/or injection of X-ray contrast in the antecubital vein, at the choice of the implanter. One or more vascular punctures will be performed, as needed.

INTERVENTIONS:
Procedure: Ultrasound guided venous access — Access of the axillary vein using ultrasound guidance.
  Arms: Ultrasound guided venous access

SUMMARY:
The study will include patients scheduled for transvenous pacemaker- or implantable defibrillator surgery, where venous access is necessary for lead implantation. A 1:1 randomization will be performed to either standard access (at the discretion of the surgeon) or ultrasound-guided using a wireless vascular transducer (Siemens Freestyle). Primary outcome is mean time to vascular access. In addition, success rate, complication rate and total procedure time will be measured.

DETAILED DESCRIPTION:
Pacemaker- and defibrillator lead implants typically involve vascular access via the left cephalic, axillar or subclavian vein. Gaining access is usually straight forward for an experienced surgeon/implanter, but can be difficult in a minority of cases, or for implanters with less experience. Complications include arterial puncture, pneumothorax and local bleeding or hematoma. Traditionally cephalic vein cut-down is the first choice, but is only available in 70% of cases, and for more complex procedures involving three electrodes, an additional access is always required.

Ultrasound guidance is very common in other vascular access areas such as femoral artery, radial artery and internal jugular vein, but has not gained widespread acceptance in pacemaker procedures. High quality studies, demonstrating superiority or non-inferiority over other access methods are lacking.

The present study will include all comer patients scheduled for transvenous pacemaker- or implantable defibrillator surgery, where venous access is necessary for lead implantation. A 1:1 randomization will be performed to either standard access (at the discretion of the surgeon) or ultrasound-guided using a wireless vascular transducer (Siemens Freestyle). Implanters with various degrees of ultrasound experience and pacemaker surgery experience will participate in the study. All implanters will receive a 2-hour training lecture and additional hands-on training for the first 3 cases, by an ultrasound-experienced anaesthesiologist.

Access time and success rate will be recorded, and all acute complications will be recorded. Primary outcome is mean time to vascular access. In addition, success rate, complication rate and total procedure time will be measured. Outcome data will be analyzed for the entire cohort, but also stratified for implanter and excluding the first 10 cases for each implanter, to compensate for various experience and individual learning curve.

ELIGIBILITY:
Inclusion Criteria:

* Planned pacemaker or implantable defibrillator surgery with at least one new transvenously placed lead.

Exclusion Criteria:

* Difficult vascular access known before surgery, where special access technique is planned or required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-02-27 (Actual); Study Completion 2025-02-27 (Actual)

PRIMARY OUTCOMES:
Mean time to complete venous access | Peroperatively
  Time from start of vascular access attempt to achieved access for the required number access points (ie number of leads)

SECONDARY OUTCOMES:
Mean time to first venous access | Peroperatively
  Time from start of vascular access attempt to achieved access for the first introducer or lead
Successrate for full venous access | Peroperatively
  Percentage of cases with achieved full venous access using the assigned technique, without having to change technique
Successrate for full venous access within 3 minutes | Peroperatively
  Percentage of cases with achieved full venous access within 3 minutes, using the assigned technique, without having to change technique
Full venous access without any complication | Peroperatively within 24 hours
  Percentage of full venous access without any complication (including arterial puncture, pneumothorax, hemothorax, local hematoma and other acute complications)

CONTACTS AND LOCATIONS:
Locations (1):
- Skane University Hospital, Lund, Sweden